CLINICAL TRIAL: NCT02232529
Title: A Two-Part Study Designed to Evaluate the Pharmacokinetic Profile of MIN-101 and Its Main Metabolites Following Single and Multiple Dose Modified Release Prototype Formulation Administration in Healthy Cytochrome P450 2D6 Extensive Metabolizer Male and Female Subjects, and to Evaluate the Relationship Between the Pharmacokinetic Profile of MIN-101 and Its Main Metabolites and Cardiovascular Parameters.
Brief Title: Pharmacokinetic Study of MIN-101 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minerva Neurosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Basic Science
Other Study IDs: MIN-101C02; 2014-001613-53 (EudraCT Number)
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia
Keywords: modified release formulation; pharmacokinetics
MeSH Terms: conditions — Schizophrenia | interventions — roluperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1: MIN-101 (Experimental): MIN-101
  modified release formulation (MR),single oral dose between 16 and 64 mg
  Interventions: Drug: MIN-101
- Part 2: MIN-101 low dose (Experimental): MIN-101
  single daily oral dose, low dose MR formulation, from Day 1 to Day 7
  Interventions: Drug: MIN-101
- Part 2: placebo (Placebo Comparator): placebo MIN-101
  daily oral dose from Day 1 to Day 7
  Interventions: Drug: Placebo
- Part 2: MIN-101 high dose (Experimental): MIN-101
  single daily oral dose, low dose MR formulation, from Day 1 to Day 7
  Interventions: Drug: MIN-101

INTERVENTIONS:
Drug: MIN-101
  Arms: Part 1: MIN-101; Part 2: MIN-101 high dose; Part 2: MIN-101 low dose
Drug: Placebo
  Arms: Part 2: placebo

SUMMARY:
The aim of the study is to assess how MIN-101 is taken up by the body when given in different amounts and in different formulations. The drug will be given as a single dose in Part 1 of the study and during Part 2 of the study as multiple dose, once daily for 7 days. The ultimate aim is to find an optimal formulation which can be developed as a once daily dose for the treatment of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males (Part 1 and Part 2) or non-pregnant, non-lactating healthy females (Part 2 only)
* Body mass index (BMI) of 18.0 to 30.0 kg/m2
* Must be CYP2D6 Extensive metabolizer
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must agree to use an adequate method of contraception

Key Exclusion Criteria:

* Subjects who have QTc > 430 in male, > 450 in female confirmed by a repeat ECG
* Any family history of sudden cardiac death and Torsade de Points
* No personal or family history of unexplained presyncope, syncope or orthostatic hypotension
* History of any drug or alcohol abuse in the past 2 years
* History or evidence of any medically diagnosed clinically significant psychiatric disorders
* Suicidal tendencies or history of suicidal attempts
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
* Females of childbearing potential who are pregnant or lactating (female subjects must have a negative urine pregnancy test at admission)
* Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
* Positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Part 1 Pharmacokinetic profile of MIN-101 and its main metabolites (AUC (0-last), Tmax, Cmax, AUC (0-inf), %AUCextrap, Lambda z, T1/2 and parent:metabolites ratio | predose and 0.5h, 1h, 1.5h, 2h, 2.5h, 3H, 4H, 6h, 8h, 10h, 12h, 14h, 16h, 20h, 24h, 48h and 72h post-dose
Part 2 - Pharmacokinetic profile of MIN-101 and its main metabolites - Absolute QT intervals and QT intervals corrected using Fridericia formula (QTcF) | predose to Day 8

SECONDARY OUTCOMES:
Part 1 Safety and tolerability (incidence of adverse events, safety laboratory, 12-lead ECGs, vital signs, physical examination) - | from predose up to 72 h post dosing
Part 1 Pharmacokinetic profile of MIN-101 in fed and fasted state | from predose up to 72 h post dosing
Part 2 Change from baseline in ECG parameters other than QT/QTc | from predose up to Day 8
  QTcB, QRS, RR, PR intervals, U waves, T waves morphology
Part 2 Change from baseline in heart rate and blood pressure | from predose up to Day 8
Part 2 Incidence of QT/QTc changes from baseline greater than 30 and 60 ms post dose | from predose up to Day 8
Part 2 Incidence of QTc values greater than 450, 480 and 500 ms post dose | from predose up to Day 8
Part 2 Safety and tolerability of MIN-101 (adverse events occurrence, physical examination, safety laboratory tests) | from predose up to Day 8

OTHER OUTCOMES:
Changes in sleep architecture and sleep continuity | Day 6

CONTACTS AND LOCATIONS:
Overall Officials: Pui Leung, M.D, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom